CLINICAL TRIAL: NCT05763368
Title: Evaluation of Proprioception in Patients With Total Hip Replacement
Acronym: PROPRIO-ATA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of participants
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Mariagrazia Benedetti, Rehabilitation Unit Head, Istituto Ortopedico Rizzoli
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 0004373
Record Dates: First submitted 2022-07-14; First posted 2023-03-10 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Coxarthrosis; Primary
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive Lateral Approach (Active Comparator)
  Interventions: Diagnostic Test: Clinical tests and proprioception evaluation
- Anterior Approach (Active Comparator)
  Interventions: Diagnostic Test: Clinical tests and proprioception evaluation

INTERVENTIONS:
Diagnostic Test: Clinical tests and proprioception evaluation — Each patient will be evaluated using clinical scales (BBS, HHS, HOOS, SF12) and ''Delos Proprioceptive System'' to assess postural stability and proprioception.

SUMMARY:
Disturbances of balance and postural stability are frequent in patients with coxarthrosis due to the damage to the mechanoreceptors, characteristic of arthritic degeneration, and muscular hypotrophy of the affected limb.

The aim of the study is to evaluate with adequate instrumentation the alterations of proprioception and postural control in patients with hip osteoarthrosis and the effectiveness of joint reconstruction in improving any deficit.

ELIGIBILITY:
Inclusion Criteria:

* Primary Osteoarthrosis
* BMI < 35 kg/m^2
* Able to stand in monopodalic support without aids / support

Exclusion Criteria:

* History of previous hip or knee replacement
* Orthopedic trauma within the previous 6 months
* Pathologies that can interfere with balance: neurological (of the central nervous system, neuropathies, movement disorders), vestibular, visual, cognitive disability, consumption of alcohol / drugs / psychoactive drugs in the 24 hours prior to the test

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline postural stability and proprioception | At baseline, 3 months, 6 months, and 12 months from surgery
  Improvement of stability, evaluated with Berg Balance Scale, 0=minimum (the worst), 56 = maximum (the best)
Change from baseline postural stability and proprioception | At baseline, 3 months, 6 months, and 12 months from surgery
  Improvement of stability and proprioception, evaluated with Delos Proprioceptive System

SECONDARY OUTCOMES:
Clinical improvements | At baseline, 3 months, 6 months, and 12 months from surgery
  Evaluation of clinical improvements using the Harris Hip Score, 0=minimum (the worst), 100 = maximum (the best)
Clinical improvements | At baseline, 3 months, 6 months, and 12 months from surgery
  Evaluation of clinical improvements using the Patient Reported Outcome Measures with HOOS (Hip disability and Osteoarthritis Outcome Score) Physical Function shortform (HOOS-PS), 0=minimum (the worst), 100 = maximum (the best)
Patient satisfaction | At baseline, 3 months, 6 months, and 12 months from surgery
  Evaluation of patient satisfaction using the 12-Item Short Form Health Survey (SF-12) 0=minimum (the worst), 100 = maximum (the best)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS-Istituto Ortopedico Rizzoli, Bologna, Italy